CLINICAL TRIAL: NCT00826488
Title: A Comparison of Breast Tomosynthesis Mammography and Conventional Breast Imaging in the Characterization of Breast Masses: A Pilot Study
Brief Title: A Comparison of Breast Tomosynthesis Mammography and Conventional Breast Imaging in the Characterization of Breast Masses
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Principal Investigator, Darlene Bird, R.T. (M), Research Coordinator, Washington University School of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: DBT11212008
Record Dates: First submitted 2009-01-20; First posted 2009-01-22 (Estimated); Last update posted 2015-06-02 (Estimated); Status verified 2015-06

CONDITIONS: Fibrocystic Disease of Breast; Breast Cancer
Keywords: Breast Cancer; Mammography; Benign masses; Breast Lump; Breast Biopsy; Breast Mass
MeSH Terms: conditions — Fibrocystic Breast Disease; Breast Neoplasms | interventions — Mammography

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- observational (Other): Observational
  Interventions: Device: Digital Breast Tomosynthesis

INTERVENTIONS:
Device: Digital Breast Tomosynthesis — Women with a positive screening mammogram called back for additional views will be asked to undergo an additional Digital Breast Tomosynthesis (3D mammogram) on the affected breast. Radiation dose is somewhat less than that of a screening mammogram.

SUMMARY:
The purpose of this study is to compare conventional breast imaging and diagnostic work-up (2 dimensional imaging) to digital breast tomosynthesis (3 dimensional imaging) in the appearance of non-calcified breast masses. It is thought that non-calcified breast masses will be better visualized with the new 3D technology.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Any race or ethnicity
* At least 35 years old
* Prior screening or full diagnostic mammogram at Barnes Jewish Breast Health Center

Exclusion Criteria:

* Unable or unwilling to undergo informed consent
* Subjects who have breast implants
* Subjects who are unable or unwilling to tolerate compression
* Subjects who are pregnant or who think they may be pregnant
* Subjects who are currently lactating
* Men
* Women less than 35 years old
* Women greater than 80 years old
* Subjects whose breasts are larger than the tomosynthesis detector

Ages: 35 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Actual)
Dates: Start 2009-03; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
It is anticipated that out of 100 subjects recalled for additional breast imaging that 10 women will be recalled for biopsy. By adding 2D & 3D imaging, it is anticipated that 30 subjects out of 100 will have needed no workup. | 9 months

CONTACTS AND LOCATIONS:
Overall Officials: Dione Farria, MD MPH, Principal Investigator — Washington University School of Medicine
Locations (1):
- JoAnne Knight Breast Center, Barnes Hospital, St Louis, Missouri, United States